CLINICAL TRIAL: NCT05232084
Title: Erector Spinae Plane Block in Different Volumes on Postoperative Pain Control Following Breast Surgery: A Randomized, Prospective Study
Brief Title: Different Volumes of Erector Spinae Plane Block for Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 26
Record Dates: First submitted 2022-01-14; First posted 2022-02-09 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Diseases
Keywords: Mastectomy and axillary dissection surgery; Postoperative pain management; Erector Spinae Plane Block
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is 30 ml volume ESPB group. The second one is 20 ml volume ESPB group
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and the anesthesiologist who will perform postoperative pain evaluation and opioid consumption will not know the group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 30 = 30 ml of Erector spinae plane block group (Active Comparator): In group 30 ml, ESPB will be performed with patients in the lateral decubitus position while the surgical site up. US probe will be placed 2-3 cm lateral to the T4 transvers process. The block needle will be inserted cranio-caudal direction and then for correction of the needle 5 ml saline will be injected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 30 ml %0.25 bupivacaine will be administered for block.
  Interventions: Drug: Bupivacaine + Fentanyl
- Group 20 = 20 ml of Erector spinae plane block group (Active Comparator): In group ESPB, ESPB will be performed with patients in the lateral decubitus position while the surgical site up. US probe will be placed 2-3 cm lateral to the T4 transvers process. The block needle will be inserted cranio-caudal direction and then for correction of the needle 5 ml saline will be injected deep into the erector spina muscle fascia. Following confirmation of the correct position of the needle 20 ml %0.25 bupivacaine will be administered for block.
  Interventions: Drug: Bupivacaine + Fentanyl

INTERVENTIONS:
Drug: Bupivacaine + Fentanyl — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol included 10 mcg bolus without infusion dose, 10 min lockout time and 4 hour limit. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.

SUMMARY:
Postoperative pain is an important issue in female patients underwent breast surgery. Postoperative effective pain treatment provides early mobilization and shorter hospital stay. The US-guided erector spina plane block (ESPB) may be used for postoperative pain treatment following breast surgery. It is a relatively novel interfascial block that was defined by Forero et al. It has been reported that ESPB provides effective analgesia management for several breast surgeries.

DETAILED DESCRIPTION:
Various methods may be performed to reduce the use of systemic opioids and for effective pain treatment following mastectomy and axillary dissection surgery. Ultrasound (US)-guided interfascial plane blocks have been used increasingly due to the advantages of ultrasound in anesthesia practice.

The US-guided erector spina plane block (ESPB) provides thoracic analgesia at T5 level and abdominal analgesia at T7-9 level. ESPB contains a local anesthetic injection into the deep fascia of erector spinae. Visualization of sonoanatomy is easy, and the spread of local anesthesic agents can be easily seen under the erector spinae muscle. Thus, analgesia occurs in several dermatomes with cephalad-caudad way. In the literature, it has been reported that ESP block provides effective analgesia after several surgeries such as open heart surgery, breast surgery, thoracoscopic and abdominal operations.

The aim of this study is to compare the efficacy of the different volumes of US-guided ESPB for postoperative analgesia after mastectomy and axillary dissection surgery. The primary aim is to compare postoperative opioid consumption, and the secondary aim is to evaluate pain scores (VAS), and adverse effects related with opioids (allergic reaction, nausea, vomiting).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-II
* Scheduled for mastectomy and axillary dissection surgery under general anesthesia

Exclusion Criteria:

* anticoagulant treatment,
* known local anesthetic allergy,
* infected skin around the block site,
* pregnancy or breast-feeding,
* back abnormalities

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients who will undergo breast surgery will be included
Enrollment: 40 (Actual)
Dates: Start 2022-01-27 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-05-25 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption (need and demand as microgram) | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The primary aim is to compare postoperative opioid (fentanyl) consumption on patient controlled analgesia device.
  The parameters on PCA devices such as delivery and demand will be assessed

SECONDARY OUTCOMES:
Pain scores (Visual analogue scores-VAS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours
  Postoperative pain assessment will be performed using the VAS score (0 = no pain, 10 = the most severe pain felt). The VAS scores will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH. Erector spinae plane block and thoracic paravertebral block for breast surgery compared to IV-morphine: A randomized controlled trial. J Clin Anesth. 2020 Feb;59:84-88. doi: 10.1016/j.jclinane.2019.06.036. Epub 2019 Jul 4. PMID 31280100
- [Background] Altiparmak B, Korkmaz Toker M, Uysal AI, Gumus Demirbilek S. Comparison of the efficacy of erector spinae plane block performed with different concentrations of bupivacaine on postoperative analgesia after mastectomy surgery: ramdomized, prospective, double blinded trial. BMC Anesthesiol. 2019 Mar 4;19(1):31. doi: 10.1186/s12871-019-0700-3. PMID 30832580
- [Background] Uda Y, Byrne K, Brahmbhatt A, Gotmaker R, Lim D, Konishi Y, Eves TK, Paxton E, Barrington MJ. A pilot randomized-controlled trial evaluating the erector spinae plane block in thoracic and breast surgery. Can J Anaesth. 2020 Oct;67(10):1371-1380. doi: 10.1007/s12630-020-01759-5. Epub 2020 Jul 21. PMID 32696226
- [Background] Sharma S, Arora S, Jafra A, Singh G. Efficacy of erector spinae plane block for postoperative analgesia in total mastectomy and axillary clearance: A randomized controlled trial. Saudi J Anaesth. 2020 Apr-Jun;14(2):186-191. doi: 10.4103/sja.SJA_625_19. Epub 2020 Mar 5. PMID 32317873